CLINICAL TRIAL: NCT05768269
Title: A Long-Term Follow-up Study for Subjects Previously Treated With A Century Therapeutics Cellular Therapy Product
Brief Title: A Study for Participants Previously Treated With Century Therapeutics Cellular Therapy Product
Status: Recruiting | Type: Observational
Sponsor: Century Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CNTY-LTFU-01
Record Dates: First submitted 2023-03-03; First posted 2023-03-14 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Hematological Malignancy; Solid Tumor Malignancy
Keywords: Century Therapeutics; Cellular Therapy; Cell therapy; Malignancy
MeSH Terms: conditions — Hematologic Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cellular Therapy: Participants who have previously received an induced pluripotent stem cell (iPSC)-derived, ex vivo genome edited cellular therapy product in an eligible Century-sponsored index trial will be enrolled in this study for up to 180 months following the last treatment with a cellular therapy product in an eligible index trial.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — As this is a non-interventional rollover, long-term safety follow-up study, no intervention will be administered.

SUMMARY:
This study is designed to collect long-term safety and survival data from participants previously treated in an eligible Century-sponsored index trial. This is an observational study, and the elements of the study design allow for important follow-up for safety, survival, and the continued evaluation of any late adverse events (AEs) that may appear after treatment with such cellular products. Additionally, collection of persistence data from participants will support the identification of any long-term risks or late AEs that may be causally related to treatment with such cellular products.

ELIGIBILITY:
Inclusion Criteria:

* Participant has provided written informed consent prior to any long-term follow-up (LTFU) study-specific procedures.
* Participants received at least one treatment with a cellular therapy product in an eligible index trial.
* Participant was withdrawn, early discontinued or completed an eligible index trial.
* Participant is willing and able to comply with scheduled visits, study plan, and other study procedures.

Exclusion Criteria:

-This study has no exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who have been previously treated with cellular therapy products in an eligible investigational index trial.
Sampling Method: Non-Probability Sample
Enrollment: 375 (Estimated)
Dates: Start 2024-04-29 (Actual); Primary Completion 2040-03 (Estimated); Study Completion 2040-03 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With any Adverse Events of Special Interest (AESI) | Up to 180 months

SECONDARY OUTCOMES:
Number of Participants With Cellular Product-related Serious Adverse Events (SAEs) | Up to 180 months
Overall Survival (OS) | From first dose of study drug up to end of the study or death whichever occurs first (up to 180 months)
  OS is defined as the time from first treatment with a cellular therapy product in the index trial to date of death by any cause.
Percentage of Participants With Persistent Product | Up to 180 months
  Persistence of the cellular product will be assessed by a droplet digital polymerase chain reaction molecular test to evaluate transgene copies in the peripheral blood. Summary of persistence sample results (positive/negative) will be reported.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - University of Southern California - Norris Comprehensive Cancer Center, Los Angeles, California
  - University of Maryland Medical Center, Baltimore, Maryland
  - Corewell Health, Grand Rapids, Michigan
  - Levine Cancer Institute, Charlotte, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Swedish Cancer Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No